CLINICAL TRIAL: NCT03122340
Title: Single-center Double-blind, Randomized, Placebo-controlled Study of the Safety and Efficacy of Polyprenols (ROPREN) in Subjects With Acute Coronary Syndrome
Brief Title: Polyprenols (Ropren) in Acute Coronary Syndrome
Acronym: POLYNCOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Evgeny V. Vyshlov, Principal investigator, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Polyprenols
Record Dates: First submitted 2017-04-06; First posted 2017-04-20 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Polyprenols; Cholesterol
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ropren; Oils

STUDY DESIGN:
Intervention Model Description: Single-center double-blind, randomized, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Oil: 8 drops 3 times per day for 3 weeks, then 5 drops 3 times per day for 5 weeks
  Interventions: Other: Oil
- Polyprenol Group (Experimental): Polyprenols (ROPREN): 8 drops 3 times per day for 3 weeks, then 5 drops 3 times per day for 5 weeks
  Interventions: Drug: Ropren

INTERVENTIONS:
Drug: Ropren — Per os 8 drops 3 times per day for 3 weeks, then 5 drops 3 times per day for 5 weeks
  Other Names: Polyprenol
  Arms: Polyprenol Group
Other: Oil — Per os 8 drops 3 times per day for 3 weeks, then 5 drops 3 times per day for 5 weeks
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
The aim of this study is to determine efficacy and safety of polyprenols (ROPREN) using in patients with acute coronary syndrome

DETAILED DESCRIPTION:
This study is randomized double blind placebo controlled. Patients with acute coronary syndrome taking standard therapy including atorvastatin 40 mg/day were randomized into 2 groups: group 1 takes Ropren 8 drops 3 times per day for 3 week, then 5 drops 3 times per day for 5 weeks; group 2 take placebo in the same dose regimen. The hepatoprotective, hypolipidemic, antiinflammatory, cognitive, antidepression functions evaluates after one and two - month therapy

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome
* Informed consent received

Exclusion Criteria:

* Patient's incapacity to take accurately drops by oneself
* Cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Сardiospecific enzymes | At 9 days after acute coronary syndrome
  The levels of CK, CK-MB, Troponin I
Hepatic enzymes | At 2 months after acute coronary syndrome
  The levels of AST, ALT, Alkaline phosphatase, Gamma glutamine transferase
Inflammatory enzymes | At 2 months after acute coronary syndrome
  CRP, Interleukin-6, products of lipid peroxidation
Cognitive Function | At 2 months after acute coronary syndrome
  Cognitive function test evolution: Montreal Cognitive Assessment Scale
Lipid spectrum | At 2 months after acute coronary syndrome
  Cholesterol, triglycerides, lipoproteins high density, lipoproteins low density
Bilirubin | At 2 months after acute coronary syndrome
  Total and direct
Cognitive Function Anxiety | At 2 months after acute coronary syndrome
  Cognitive function test evolution: Sheehan Anxiety Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Popov, MD, PhD, Study Director — Tomsk NRMC
Locations (1):
- Cardiology Research Institute, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vyshlov EV, Tsoy EI, Sultanov VS, Trusov VB, Ryabov VV. Hypolipidemic and Hepatoprotective Effects of a Polyprenol-Containing Drug in Patients with Acute Coronary Syndrome. Bull Exp Biol Med. 2018 Jul;165(3):319-321. doi: 10.1007/s10517-018-4159-x. Epub 2018 Jul 12. PMID 29998439